CLINICAL TRIAL: NCT04636905
Title: Evaluation of the Survivorship Wellness Group Program: An Interdisciplinary Goal-Setting Clinical Group Program for Survivors of Cancer at UCSF
Brief Title: Evaluation of Survivorship Wellness Group Program for Patients Treated at University of California, San Francisco (UCSF)
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 20802
Record Dates: First submitted 2020-11-13; First posted 2020-11-19 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Cancer
Keywords: Quality of Life; Survivorship; Health Behaviors
MeSH Terms: conditions — Neoplasms; Health Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Survivorship Wellness Group: Participants will be enrolled in a 15 week program to assess quality of life and general health outcomes
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Participants will be asked to complete a series of questionnaires assessing quality of life and other general health outcomes

SUMMARY:
Interdisciplinary psychological interventions targeting survivorship are not only understudied but face several implementation challenges. For this project, the study team is proposing to analyze these data to report on preliminary pilot outcomes, as well as acceptability and feasibility of the implementation of the Survivorship Wellness Group Program, an interdisciplinary wellness and health-behavior change program for survivors of cancer, who have completed treatment at University of California, San Francisco and are currently without evidence of active disease.

DETAILED DESCRIPTION:
STUDY OBJECTIVES:

1. To examine the feasibility and acceptability of implementing an interdisciplinary goal-setting clinical group program focused on domains of physical, psychological, and spiritual wellness for survivors of cancer at University of California, San Francisco.
2. To determine preliminary efficacy of the Survivorship Wellness intervention in regards to:

   1. Increasing knowledge of and perceived confidence in execution of health behavior changes in domains of physical, emotional, and spiritual wellness for survivors of cancer
   2. Increasing quality of life
   3. Reducing symptoms of depression and anxiety
   4. Increasing physical activity

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Treated for any kind of cancer at University of California, San Francisco, though finished with active treatments (defined as chemotherapy, radiation, or surgery) at time of enrollment, and without evidence of current active cancer
* Sufficient cognitive ability to participate in group activities as determined by their attending medical oncologist or surgeon

Exclusion Criteria:

* Non-English speaking
* Primary cancer treatment outside of UCSF
* Currently receiving non-maintenance therapies (chemotherapy or radiation) for active cancer
* Psychiatric illness that would affect the ability to participate in a group activity

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Survivors of cancer who have been treated at University of California, San Francisco
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Change in the Patient Reported Outcome Measurement Information System (PROMIS) Depression Short Form Depression scores over time | Up to 16 weeks
  The PROMIS Depression Short form consists of 4 items addressing patient depression with item response scores ranging from 1 (never) to 5 (Always). Raw scores are converted to scaled T-scores with higher scores indicating a greater level of depression.
Changes in the Patient Reported Outcome Measurement Information System (PROMIS) Anxiety Short Form scores over time | Up to 16 weeks
  The PROMIS Anxiety Short form consists of 2 items addressing patient anxiety with item response scores ranging from 1 (never) to 5 (Always). Raw scores are converted to scaled T-scores with higher scores indicating a greater level of anxiety.
Changes in the Functional Assessment of Cancer Therapy scale (FACT-G) scores over time | Up to 16 weeks
  The FACT-G is a 27-item questionnaire designed to measure four domains of health related quality of life (HRQOL) in cancer patients with 4 domains of interest: Physical, social, emotional, and functional well-being. Each tem response score ranges from 0 (not at all) to 5 (very much). The total score is a sum of the subscale scores, with a range from 0 - 108. The higher the score, the better the HRQOL.
Frequency of participant responses to Program Satisfaction survey item | Week 16
  Program satisfaction is measured by the participant's response to the following item: "How satisfied were you, overall, with this program?". Responses ranged from Not at all satisfied, Somewhat satisfied, Mostly satisfied, and Extremely satisfied. Responses will be counted and reported by category.
Changes in the frequency of participant responses cancer survivorship wellness survey: Importance | Up to 16 weeks
  The 16 item cancer survivorship wellness survey assesses each participant for their level of importance in learning about various wellness topics of cancer survivorship and their current knowledge of these topics. Each item addressing importance is rated by the participant in terms of how important it is to learn about topics specific to cancer survivorship. Items are rated according to 5 categories "Not at all important", "Somewhat important", "Moderately important", "Very important", and "Extremely important".
Changes in the frequency of participant responses cancer survivorship wellness survey- Knowledge | Up to 16 weeks
  The 16 item cancer survivorship wellness survey assesses each participant for their level of importance in learning about various wellness topics of cancer survivorship and their current knowledge of these topics. Each item addressing knowledge is rated by the participant in terms of how knowledgeable the participants are regarding topics specific to cancer survivorship. Items are rated according to 5 categories "Not at all knowledgeable", "Somewhat knowledgeable", "Moderately knowledgeable", "Very knowledgeable", and "Extremely knowledgeable".
Changes in the frequency of participant responses to exercise frequency survey item | Up to 16 weeks
  The frequency of current exercise for participants was measured by a single item "How frequently do you exercise currently"? Responses are comprised of 5 categories: "Every day", "Several times per week", "Once per week", "Less than once per week", "Several times per month", "Once per month", and "Less than once per month"
Changes in the frequency of participant responses to exercise intensity survey item | Up to 16 weeks
  The intensity of current exercise for participants was measured by a single item "How would you rate the intensity of your current exercise regimen?". Responses are comprised of 5 categories: "Very low intensity", "Light intensity", "Moderate intensity", and "High intensity".

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Chesney, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No